CLINICAL TRIAL: NCT03254147
Title: Medical Need of Oral Anti-coagulant Reversal in Japan: Epidemiological Assessment of Head Trauma, Fracture, and Emergency Surgery Using Large Scale Claims Database (Please Note That This Study Contains no Patients Treated With Idarucizumab Although the Study Number Begins With 1321; the Study Contains Only Patients Treated With OACs, Namely Warfarin, Dabigatran, Edoxaban, Apixaban, Rivaroxaban, Edoxaban)
Brief Title: Medical Need of OAC Reversal
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1321-0022
Record Dates: First submitted 2017-08-17; First posted 2017-08-18 (Actual); Results first posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin; Dabigatran; apixaban; edoxaban; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients prescribed with Oral Anti-coagulants: warfarin and non-vitamin K dependent oral anti-coagulants
  Interventions: Drug: warfarin; Drug: dabigatran; Drug: Apixaban; Drug: Edoxaban; Drug: Rivaroxaban

INTERVENTIONS:
Drug: warfarin — warfarin
Drug: dabigatran — Non-vitamin K dependent oral anti-coagulants (NOACs)
  Other Names: PRADAXA, PRAZAXA
Drug: Apixaban — Non-vitamin K dependent oral anti-coagulants (NOACs)
Drug: Edoxaban — Non-vitamin K dependent oral anti-coagulants (NOACs)
Drug: Rivaroxaban — Non-vitamin K dependent oral anti-coagulants (NOACs)

SUMMARY:
This is a retrospective, observational, claims cohort study to assess, for adult patients initiating an oral anticoagulant for NVAF

DETAILED DESCRIPTION:
This is a retrospective, observational, claims cohort study to assess, for adult patients initiating an oral anticoagulant for NVAF, the incidence rates of emergency surgery, major bleeding due to trauma, and major bleeding due to fracture, overall and stratified by age (<64, 65-74, >75). The secondary objective is to estimate the overall and age stratified incidence of cardiac tamponade and peri-cardiocentesis.

ELIGIBILITY:
Inclusion Criteria:

->18 year old non-valvular atrial fibrillation (NVAF) patients

* Prescribed dabigatran, rivaroxaban, apixaban, edoxaban or warfarin
* Patients with confirmed date of initiation of OACs
* Patients with a minimum of 6 months of enrolment data prior to index date
* Has an index date between 14th of March 2011 to 30 June, 2016

Exclusion Criteria:

* Patients receiving two or more oral anti-coagulants at the same time at index date
* Patients with prescriptions of index treatment in the 6 months prior to index date
* Patients without enrolment period of at least six month in the database

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients with atrial fibrillation contained in the Medical Data Vision (MDV) database which is a Japanese, nationwide claims data containing approximately 16 million patients cumulatively. The data cut is between March 2011 to June 2016, and the patients in the MDV database are those who have visited DPC hospitals (diagnostic procedure combination, a lump-sum payment system based on disease diagnosis to be treated similar to Medicare/Medicaid in the USA) hospitals which provide acute in-patient, as well as outpatient care.
Sampling Method: Non-Probability Sample
Enrollment: 53969 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yasaka M, Yokota H, Suzuki M, Yamane T, Ono Y. Incidence Rates of Bleeding and Emergency Surgery Due to Trauma or Fracture Among Japanese Patients with Non-valvular Atrial Fibrillation Receiving Oral Anticoagulation Therapy. Cardiol Ther. 2020 Jun;9(1):189-199. doi: 10.1007/s40119-020-00171-w. Epub 2020 May 11. PMID 32394292

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-interventional study based on existing health insurance claims data
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients met all strictly implemented inclusion/exclusion criteria. Patients were not to be entered to trial if any one of the specific entry criteria was violated.
Groups:
- Patients Prescribed With Non-warfarin Oral Anti Coagulants: Patients prescribed with Non-warfarin Oral Anti Coagulants (NOACs) (dabigatran, rivaroxaban, apixaban, edoxaban) or warfarin were grouped as a single exposure group and analysed as a whole. On treatment duration was expressed in patient year for the follow-up duration to calculate the incidence of various clinical events during the on-treatment duration.
Period: Overall Study
Arm/Group | Patients Prescribed With Non-warfarin Oral Anti Coagulants
Started | 53969 (The number of patients meeting the inclusion and exclusion criteria)
Completed | 53969
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are based on the number of patients meeting the inclusion and exclusion criteria.
Arm/Group | Patients Prescribed With Non-warfarin Oral Anti Coagulants
Number analyzed (Participants) | 53969
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Baseline characteristics are based on the number of patients meeting the inclusion and exclusion criteria.
  Years | 76 (10)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics are based on the number of patients meeting the inclusion and exclusion criteria.
  Participants
    Female | 21587
    Male | 32382
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics are based on the number of patients meeting the inclusion and exclusion criteria.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 53969
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics are based on the number of patients meeting the inclusion and exclusion criteria.
  Participants
    American Indian or Alaska Native | 0
    Asian | 53969
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Emergency Surgery and Major Bleeding Due to Fracture or Trauma.
Description: The number of patients with emergency surgery and major bleeding due to fracture or trauma. Where emergency surgery defined as any surgical procedure (International Classification of Diseases (ICD) 10 code K000-879) performed on the same day as hospital admission with additional claims, major bleeding due to fracture is any bleeding associated with hospitalization or blood transfusion (ICD10 code E83.111) accompanied by any fracture, and major bleeding due to trauma is any bleeding associated with hospitalization or blood transfusion (ICD10 code E83.111) accompanied by any trauma.
Time Frame: One year
Population: Results are based on the number of patients meeting the inclusion and exclusion criteria.
Measure: Number; unit: Number of Patients
Arm/Group | Patients Prescribed With Non-warfarin Oral Anti Coagulants
Number analyzed (Participants) | 53969
Number of Patients
  Age <=64: number analyzed (Participants) | 6960
  Age <=64 | 14
  Age 65-74: number analyzed (Participants) | 14568
  Age 65-74 | 35
  Age >=75: number analyzed (Participants) | 32441
  Age >=75 | 84

2. Secondary Outcome: The Number of Patients With Cardiac Tamponade and Pericardiocentesis.
Description: The number of patients with cardiac tamponade and pericardiocentesis. Cardiac tamponade diagnosis (ICD 10 code 4200001) on the same or next day as catheter ablation or percutaneous coronary intervention (PCI), Pericardiocentesis (Medical Data Vision (MDV) procedure code 140010510) on the same or next day as catheter ablation or PCI.
Time Frame: One year
Population: Results are based on the number of patients meeting the inclusion and exclusion criteria.
Measure: Number; unit: Number of Patients
Arm/Group | Patients Prescribed With Non-warfarin Oral Anti Coagulants
Number analyzed (Participants) | 53969
Number of Patients | 1

ADVERSE EVENTS:
Time Frame: No adverse event reporting was done.
Description: This is a cohort study based on existing data; therefore, it is not feasible to make a causality assessment at the individual case level. Hence no adverse event reporting was done.
Arm/Group | Patients Prescribed With Non-warfarin Oral Anti Coagulants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The findings from this study may not be generalizable to other Japanese population outside of Diagnosis Procedure Combination (DPC) hospitals. All information of each patient is from consent giving DPC hospitals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT03254147/Prot_SAP_000.pdf